CLINICAL TRIAL: NCT03388385
Title: The Effects of a Single Intravenous Iron Upon Vascular Endothelium and Some Parameters of Oxidative Stress in Patients With Non-dialysis Chronic Kidney Disease
Brief Title: Acute Effects of Intravenous Iron on Oxidative Stress and Endothelial Dysfunction in Non-dialysis CKD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Carol Davila University of Medicine and Pharmacy (Other)
Collaborators: S.C. Sanador S.R.L (Other)
Responsible Party: Principal Investigator, Ana-Maria Mehedinti, Teaching Assistent, Carol Davila University of Medicine and Pharmacy
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 10488/19.04.2016
Record Dates: First submitted 2017-12-18; First posted 2018-01-03 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Renal Anemia; Iron Toxicity; Oxidative Stress; Endothelial Dysfunction
Keywords: CKD, anemia, iron, endothelial dysfunction, oxidative stress
MeSH Terms: conditions — Anemia | interventions — Sodium Chloride; ferric carboxymaltose

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Intervention: 250 mL Sodium Chloride 0.9% Intravenous Solution, representing control infusion, over 30 minutes.
  Interventions: Drug: Sodium Chloride 0.9% Intravenous Solution; Drug: Ferinject
- Ferric carboxymaltose (Active Comparator): Intervention: 1000 mg Ferinject in 250 mL 0.9%NaCl, representing medication in study infusion, over 30 minutes.
  Interventions: Drug: Sodium Chloride 0.9% Intravenous Solution; Drug: Ferinject

INTERVENTIONS:
Drug: Sodium Chloride 0.9% Intravenous Solution — Physiologic saline infusion will be infused in day 1.
  Other Names: Physiologic saline
Drug: Ferinject — Ferric carboxymaltose will be infused in day 2.
  Other Names: Ferric carboxymaltose

SUMMARY:
The purpose of this study is to investigate the effects of acute intravenous iron administration on the endothelial function in non-dialysis Chronic Kidney Disease stages G3-G5 patients with anemia and iron deficiency, in relation to changes in oxidative and nitrosative status.

ELIGIBILITY:
Inclusion Criteria:

* Chronic kidney disease stages G3-G5 (defined according to KDIGO criteria);
* Anemia (defined according to KDIGO criteria) and iron deficiency defined as serum ferritin < 100 ng/mL and/or TSAT < 20% (KDIGO).

Exclusion Criteria:

* contraindications of intravenous iron therapy: iron allergy, active infection, hemochromatosis, iron overload (serum ferritin > 500 ng/mL and/or transferrin saturation > 50%);
* treatment with iron and erythropoiesis-stimulating agents (at the time of recruitment and 6 months previously);
* active smoker status;
* antioxidant food supplements treatment in the last 3 months;
* clinically manifest bleeding;
* another cause of anemia (hemoglobinopathies, vitamin B12 and/or folic acid deficiency suggested by the megaloblastic peripheral blood smears's appearance, multiple myeloma and other paraproteinemias);
* severe anemia (Hb < 7 g/dl);
* baseline FMD < 7% (the existence of atherosclerosis which limits arterial reactivity);
* cancer (currently or in the past 6 months);
* hepatopathies (increased serum transaminases ≥ 3 x normal value) or hepatic impairment ≥ grade Child B;
* autoimmune disorders or significant inflammation (as defined by C-reactive protein > 5 mg/L);
* pregnancy or lactation;
* participation in other clinical trials over the upast 3 months;
* patient unwillingness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2022-12-20 (Estimated)

PRIMARY OUTCOMES:
Effect on endothelial function | through study completion, an average of 1 year
  Description of the endothelial function variation (changing in flow-mediated vasodilatation (FMD) endothelium-dependent, and also in serum sICAM-1, sVCAM-1 and nitric oxide metabolism parameters ) after administration of a single intravenous dose of iron versus a control solution, in CKD non-dialysis patients.
Oxidative stress | through study completion, an average of 1 year
  Description of some free radicals production's markers (lipid peroxidation and carbonyl stress assessment) and in antioxidant system in plasma markers variation after administration of a single intravenous iron dose versus a control solution, in non-dialysis CKD subjects.

SECONDARY OUTCOMES:
Correlation between endothelial dysfunction and oxidative stress markers | through study completion, an average of 1 year
  Evaluation of correlations between changes in oxidative stress parameters and endothelial function after a single intravenous iron administration compared to a control solution in non-dialysis CKD subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Mircescu, Professor, Study Chair — Carol Davila University of Medicine and Pharmacy; Cristina Capusa, Assoc. Prof., Study Director — Carol Davila University of Medicine and Pharmacy
Locations (1):
- "Dr. Carol Davila" Teaching Hospital of Nephrology, Bucharest, Romania